CLINICAL TRIAL: NCT00492674
Title: The Effect of Perioperative Neuromuscular Training on the Outcome of Total Knee Arthroplasty: A Double Blind Randomized Prospective Study
Brief Title: The Effect of Perioperative Neuromuscular Training on the Outcome of Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35/07
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-04

CONDITIONS: Knee Osteoarthritis
Keywords: TKA; Arthroplasty; Knee; Osteoarthritis; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: APOS biomechanical gait system
Procedure: Physical Therapy

SUMMARY:
Introduction: Total knee arthroplasty (TKA) is a consensus treatment for end-stage knee osteoarthritis. The peri-operative rehabilitation is an important part of the outcome of such procedure. Previous studies have shown that there is correlation between both pre-operative functional status and the intensiveness of the post-operative rehabilitation to the post operative function of the patient.

An important part of the peri-operative rehabilitation in TKA is the neuromuscular control re-education.

A novel biomechanical device comprising of four individually calibrated elements attached onto foot-worn platforms was recently developed. This device is capable of bringing the patient to a functional bio-mechanical alignment during standing and walking, while simultaneously strengthening dynamic stabilizers and training neuromuscular control by means of controlled biomechanical perturbations.

Objectives: The aim of this study is to evaluate the influence of pre and post operative training with the biomechanical device mentioned above on the functional outcome and quality of life of patients undergoing TKA.

Design and Setting: Randomized, controlled and double blind prospective trial

Patients: 120 patients who are candidates to TKA

Interventions: Patients will randomly assigned into five groups (active, sham and control) and will followed for fourteen months (two moths pre-operative and twelve months post-operative). All groups will undergo post-operative physical therapy (PT) according to the standard guidelines. In addition, the active groups will be treated with the device and its four biomechanical elements that had been individually calibrated for each patient. The sham group will be treated with the same device; however, the biomechanical elements will have zero perturbation and will be positioned along the central longitudinal line of the shoe-platform. The control group will be treated only according to the standard post-operative protocol.

The five groups:

1. Pre- operative BD training and post-operative PT and BD training
2. Pre- operative sham training and post-operative PT and BD training
3. Pre- operative sham training and post-operative PT and sham training
4. No pre-operative training (according to the guidelines in Israel) and post-operative PT and BD training.
5. No pre-operative training (according to the guidelines in Israel) and post-operative PT and sham training.

Primary Outcome Measures: Spatio-temporal measures (recorded by Gait-Rite™) and the Aggregated Locomotor Function (ALF) assessment.

Secondary Outcome Measures: Pain and function questionnaire measured by the Western Ontario and McMaster Osteoarthritis Index (WOMAC) and Quality of life will be evaluated by the SF-36 quality of life questionnaire.

Measurements will be taken at day-1 (two months before the TKA) and at four more stations: 1 Week prior to the TKA, Three months post the TKA, six months post the TKA and twelve months post the TKA

DETAILED DESCRIPTION:
Introduction: Total knee arthroplasty (TKA) is a consensus treatment for end-stage knee osteoarthritis. The peri-operative rehabilitation is an important part of the outcome of such procedure. Previous studies have shown that there is correlation between both pre-operative functional status and the intensiveness of the post-operative rehabilitation to the post operative function of the patient.

An important part of the peri-operative rehabilitation in TKA is the neuromuscular control re-education.

A novel biomechanical device comprising of four individually calibrated elements attached onto foot-worn platforms was recently developed. This device is capable of bringing the patient to a functional bio-mechanical alignment during standing and walking, while simultaneously strengthening dynamic stabilizers and training neuromuscular control by means of controlled biomechanical perturbations.

Objectives: The aim of this study is to evaluate the influence of pre and post operative training with the biomechanical device mentioned above on the functional outcome and quality of life of patients undergoing TKA.

Design and Setting: Randomized, controlled and double blind prospective trial

Patients: 120 patients who are candidates to TKA

Interventions: Patients will randomly assigned into five groups (active, sham and control) and will followed for fourteen months (two moths pre-operative and twelve months post-operative). All groups will undergo post-operative physical therapy (PT) according to the standard guidelines. In addition, the active groups will be treated with the device and its four biomechanical elements that had been individually calibrated for each patient. The sham group will be treated with the same device; however, the biomechanical elements will have zero perturbation and will be positioned along the central longitudinal line of the shoe-platform. The control group will be treated only according to the standard post-operative protocol.

The five groups:

1. Pre- operative BD training and post-operative PT and BD training
2. Pre- operative sham training and post-operative PT and BD training
3. Pre- operative sham training and post-operative PT and sham training
4. No pre-operative training (according to the guidelines in Israel) and post-operative PT and BD training.
5. No pre-operative training (according to the guidelines in Israel) and post-operative PT and sham training.

Primary Outcome Measures: Spatio-temporal measures (recorded by Gait-Rite™) and the Aggregated Locomotor Function (ALF) assessment.

Secondary Outcome Measures: Pain and function questionnaire measured by the Western Ontario and McMaster Osteoarthritis Index (WOMAC) and Quality of life will be evaluated by the SF-36 quality of life questionnaire.

Measurements will be taken at day-1 (two months before the TKA) and at four more stations: 1 Week prior to the TKA, Three months post the TKA, six months post the TKA and twelve months post the TKA

ELIGIBILITY:
Inclusion Criteria:

* Candidates for total knee arthroplasty (d/t osteoarthritis)
* All operated by the same Surgeons (Prof. Nahum Halperin's group)
* Identical kind of Prosthesis in use (zimmer Lps-Flex Mobile)

Exclusion Criteria:

* Prior joint arthroplasty
* A pathology in additional segment (ankle, hip)
* Other muscular or neurological disease/condition
* Mentally or physically impairment that will prevent the patinet from proper use of the biomechanical device.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nahum Halperin, MD, Principal Investigator — Asaf-Harofeh Medical Center; Zeevi Dvir, PhD, Study Chair — Tel Aviv University; Noga Gal, Msc, Principal Investigator — Tel Aviv University